CLINICAL TRIAL: NCT05075694
Title: the Effect of Therapeutic Touch on Sleep Quality and Fatigue in Menopausal Women
Brief Title: Cukurova University Faculty of Medicine Non-interventional Clinical Research Institutional Ethics Committe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ozlem Yalcinkaya, Msc Student, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.07.2021/46
Record Dates: First submitted 2021-09-16; First posted 2021-10-13 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Menopause; Sleep; Fatigue; Therapeutic Touch
Keywords: Menopause; Sleep; Fatigue; Therapeutic touch
MeSH Terms: conditions — Fatigue | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: This study was conducted as a parallel randomized-controlled, single-blind, single-centered, interventional study with a pre-test and post-test design
Who Masked: Participant
Masking Description: In this study, while the intervention group was administered Therapeutic Touch , the control group was administered Sham Therapeutic Touch (STT). The interventions in the study were implemented using the literature information as well as the Therapeutic Touch Practice Procedure (TTPP) and Sham Therapeutic Practice Procedure (STPP). To administer the TT practice, the researcher received a certificate by participating in the first and second-level courses held by the International Therapeutic Touch Association.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Therapeutic touch (TT) is a treatment that takes an average of 15-20 min, in which energy in the universe is transferred through the hands of the practitioner to eliminate the imbalance in the individual's energy field and facilitate healing. The intervention group (TT group) received therapeutic touch for 10 minutes a day for five consecutive days. The practice was implemented in line with Therapeutic Practice Procedure.
  Interventions: Behavioral: Therapeutic Touch
- Control (Sham Comparator): Placebo: Sham Therapeutic Touch (STT) The control group was administered STT instead of TT for 10 minutes for successive 5 days. The practice was implemented in line with Sham Therapeutic Touch Practice Procedure (STTPP).
  Interventions: Other: Sham Therapeutic Touch

INTERVENTIONS:
Behavioral: Therapeutic Touch — Therapeutic Touch performed in line with the Therapeutic Touch Practice Procedure included the following steps: centering, assessing, rebalancing, reassessing, reexamining, grounding, and closure.
  Arms: Experiment
Other: Sham Therapeutic Touch — The control group was administered STT instead of TT for 10 minutes for successive 5 days. The practice was implemented in line with STTPP. The practice was implemented by not centering or intending to help to heal, by moving at a longer distance, and by imitating the TT practice protocol visually.
  Arms: Control

SUMMARY:
This research was carried out to determine the effect of therapeutic touch on sleep quality and fatigue in menopausal women.

DETAILED DESCRIPTION:
Methods: This randomized controlled experimental study was conducted with 48 (24 in the intervention group and 24 in the control group) women who sought treatment in the gynecological outpatient clinic of a public hospital. According to the study procedure, while the intervention group received therapeutic touch, the control group received SHAM therapeutic touch for 10 minutes a day for five consecutive days. Data were collected through the Personal Information Form, the Pittsburgh Sleep Quality Index, and the Piper Fatigue Scale.

Results: The median post-test total sleep quality score was significantly lower in the intervention group than in the control group (p=0.010). However, the mean total fatigue scores did not differ significantly between the groups (p=0.917).

Conclusions: The results of this study showed that therapeutic touch was effective in improving sleep quality, but it did not affect fatigue in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

The study included women who agreed to participate in the study, lived in the city center, were at least literate, were in the natural premenopausal (irregular menstrual cycle within the last three months), perimenopausal (amenorrhea for 3-11 months or increased irregular menstruation), or postmenopausal (amenorrhea for more than 12 months) periods, were open to communication and cooperation, and could speak Turkish.

Exclusion Criteria:

The women who received hormone replacement treatment, used drugs for sleep problems and depression, were diagnosed with a medical psychiatric disease, and had sensitivity or problems about touching were excluded.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | 9 months
  The Turkish version of the Pittsburgh Sleep Quality Index (PSQI), which was developed by Buyssee et al. (1989), was used for the assessment of sleep quality. It is a self-report scale that makes a quantitative assessment of sleep quality and sleep disorders over a one-month time interval [30]. Turkish reliability and validity of the scale were performed by Ağargün et al. in our country (1996) [31]. The scale is composed of 18 items and seven sub-scales, which include Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorders, Use of Sleeping Drugs, and Daytime Dysfunction. Each item is scored between 0 and 3. The total score of the seven sub-scales gives the PSQI score. Scores to be obtained from the scale range between 0 and 21. A total score greater than 5 indicates "poor sleep quality." Cronbach's alpha reliability coefficient of the PSQI was reported 0,804 in the Turkish adaptation of the scale [31].
Fatigue | 9 months
  The Turkish version of the Piper Fatigue Scale (PFS) was utilized to assess fatigue. PFS was developed by Barbara F. Piper et al. in 1987 [32]. Turkish reliability and validity of the scale were performed by Can et al. (2001) [33]. The scale responded on a 5-point Likert scale has 22 items and four sub-scales and it aims to assess individuals' subjective perceptions about fatigue. The sub-scales are Behavioral/Severity, Affective Meaning, Sensory, and Cognitive /Mood. Calculation of the sub-scale scores is done by summing all the items in that sub-scale and dividing it by the number of items. Higher scores indicate higher fatigue levels. Total Cronbach's alpha value was reported to be 0,99 in the Turkish reliability and validity of the scale [33].

CONTACTS AND LOCATIONS:
Overall Officials: Ebru GOZUYESIL, PhD, Study Chair — Cukurova University
Locations (1):
- Ozlem Yalcinkaya, Adana, Saricam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No